CLINICAL TRIAL: NCT04649099
Title: The Leaflex™ Standalone Study Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated after completion of the Exploratory phase due to reprioritization of attention and resources by Sponsor.
Sponsor: Pi-cardia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02-CLN-019
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: The study includes two stages:
  * Exploratory stage - an exploratory examination of patients with an aim to streamline the study procedures, to reach a safe and consistent result, to evaluate the target patient population and adapt scoring protocol to optimize efficacy of the Leaflex™ procedure. The protocol does not include a formal staticstical analysis of the results of subjects enrolled in this stage.
  * Confirmatory - confirmatory analysis with an aim to demonstrate the Leaflex™ safety and performance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leaflex™ Performer (Experimental)
  Interventions: Device: Leaflex™ Performer

INTERVENTIONS:
Device: Leaflex™ Performer — A transfemoral catheter designed to treat calcific aortic stenosis by scoring the calcification in the aortic valve leaflets.

SUMMARY:
A prospective, multicenter, single-arm study aimed to assess safety and performance of the Leaflex™ Performer in the treatment of patients with symptomatic, severe aortic stenosis.

Subjects will be seen at pre- and post procedure, discharge, 30 days and at 3, 6, 9 and 12 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptomatic, severe aortic stenosis who are not recommended by the heart team for immediate treatment with surgical or transcatheter aortic valve replacement.
* Patient is willing to comply with scheduled visits and tests and is able and willing to provide informed consent.

Exclusion Criteria:

* Moderate or greater aortic regurgitation.
* Anatomic contraindications.
* Coronary, carotid, or vertebral artery disease that, in the opinion of the heart team, should be treated; or treatment of coronary artery disease ≤ 1 month prior to index procedure.
* Aortic balloon valvuloplasty ≤ 3 months prior to index procedure.
* Stroke ≤ 12 months prior to index procedure.
* History of a myocardial infarction ≤ 6 weeks prior to index procedure.
* Patients with clinically significant abnormality in cell blood count, history of bleeding diathesis or coagulopathy.
* Hemodynamic instability.
* Hypertrophic cardiomyopathy with obstruction.
* Left ventricle ejection fraction <30%.
* Ongoing severe infection, including endocarditis, or sepsis.
* Life expectancy ≤ 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Change in aortic valve area | Baseline to 3 days
  assessed by echo

SECONDARY OUTCOMES:
Rate of all-cause mortality and all-cause stroke (VARC 2) | 30 days post procedure
  Composite
Rate of worsening of aortic regurgitation | Baseline to 30 days
  by greater than 1 grade
Rate of device related adverse events | 12 months
Change in 6 minute walk test | 1, 6 and 12 months
  distance (meters)
Quality of Life Improvement | 1, 6 and 12 months
  KCCQ
Quality of Life Improvement | 1, 6 and 12 months
  EQ5D
Change in aortic valve area | 30 days, 3, 6, 9 and 12 months
  assessed by echo
Change in pressure gradients | 30 days, 3, 6, 9 and 12 months
  assessed by echo

CONTACTS AND LOCATIONS:
Locations (1):
- Gottsegen Gyorgy Hungarian Institute of Cardiology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No